CLINICAL TRIAL: NCT05391061
Title: Post Marketing Surveillance (PMS) Study for Cibinqo Tablet (Abrocitinib) in Patients With Moderate to Severe Atopic Dermatitis (AD) in Korea
Brief Title: A Study to Learn About the Study Medicine (Called Cibinqo) in People With Atopic Dermatitis
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7451074
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic Dermatitis, Abrocitinib, Cibinqo
MeSH Terms: conditions — Dermatitis, Atopic | interventions — abrocitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: Abrocitinib — Tablets
  Other Names: Cibinqo

SUMMARY:
The purpose of this non-interventional study is to learn about the safety and effectivness of Cibinqo Tablet for the possible treatment of atopic dermatitis (AD).

AD is a long-lasting itchy red rash, caused by a skin reaction.

This study is seeking participants who:

1. Are patients with moderate to severe AD who have been waiting to start treatment with Cibinqo
2. Have evidence of a personally signed and dated informed consent document indicating that the patient or their parent(s) or legal guardian, have been informed of all important details of the study Investigators will collect and record the information on each participant's experiences with Cibinqo. This study medicine is a tablet which is taken by mouth. Participants will be observed for about a year. During this time, we will study the experiences of people receiving the study medicine to help us decide if the study medicine is safe and effective.

DETAILED DESCRIPTION:
This study is a single country, multicenter, prospective, non-interventional, observational post marketing surveillance study to evaluate the safety and effectiveness of Cibinqo® Tablet in participants with moderate to severe AD in routine clinical practice in Korea.

The purpose of this study is to evaluate the safety and effectiveness of Cibinqo® Tablet in routine clinical practice for approved indications in Korea.

The study population for this study is participants 12 years of age and older who have been diagnosed with moderate to severe AD and are determined to be treated with Cibinqo® Tablet according to the approved indications in routine clinical practice in Korea.

About 3000 participants will be enrolled in several centers in this study. Pfizer Pharmaceuticals Korea will conclude a post-marketing surveillance agreement with an investigator site before performing the study.

Each investigator will sequentially enroll all subjects to whom Cibinqo is prescribed for the first time according to the "Dosage and Administration" of the approved labeling and who agree to participate in this study by signing the data privacy statement used in place of the informed consent form until the total requested cases per center are collected for this study.

There is no mandatory fixed visit schedule. The investigator will collect patient data and record the information on each patient's case report form (CRF).

ELIGIBILITY:
This study is seeking participants who should meet the usual prescribing criteria for Cibinqo® Tablets as per the Local Product Document (LPD) and should be entered into the study at the physician's discretion.

Inclusion Criteria:

1. Patients with moderate to severe AD who have been determined to start treatment with Cibinqo Tablet according to the approved indications of the medicinal product.

   • Atopic Dermatitis Cibinqo Tablet is indicated for the treatment of patients 12 years of age and older with moderate-to-severe atopic dermatitis who have required systemic therapies.
2. Evidence of a personally signed and dated informed consent document indicating that the patient or their parent(s)/legal guardian, if applicable, have been informed of all pertinent aspects of the study

Exclusion Criteria:

1. Patients who have previously received Cibinqo Tablet
2. Patients concurrently participating in other studies involving therapeutic interventions and/or investigational products
3. Patients who have contraindications to Cibinqo Tablet as specified in the approved LPD • Contraindications to Cibinqo Tablet

   * Patients with platelet count <150 × 103/mm3, an absolute neutrophil count (ANC) <1 × 103/mm3, an absolute lymphocyte count (ALC) <0.5 × 103/mm3 or who have a haemoglobin value <8 g/dL
   * Hypersensitivity to the active substance or to any of the excipients
   * Active serious systemic infetions, including tuberculosis(TB)
   * Severe hepatic impairment
   * Pregnancy and breast-feeding
   * Patients with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population for this study is patients 12 years of age and older who have been diagnosed with moderate to severe Atopic Dermatitis (AD) and are determined to be treated with Cibinqo® Tablet according to the approved indications in routine clinical practice in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2023-01-07 (Actual); Primary Completion 2027-11-22 (Estimated); Study Completion 2027-11-22 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AE's) according to frequency | Up to 52 weeks from the time of first treatment
Number of participants with Adverse Drug Reactions (ADR's) according to frequency | up to 52 weeks from the time of first treatment
Number of participants with unexpected AE's according to frequency | up to 52 weeks from the time of first treatment
Number of participants with unexpected ADR's according to frequency | up to 52 weeks from the time of first treatment
Number of participants with Serious Adverse Events (SAE's) according to frequency | up to 52 weeks from the time of first treatment
Number of participants with Serious Adverse Drug Reactions (SADR's) according to frequency | up to 52 weeks from the time of first treatment
Number of participants with Adverse Events of Special Interest (AESI) according to frequency | up to 52 weeks from the time of first treatment

SECONDARY OUTCOMES:
Proportion of participants achieving the Investigator's Global Assessment (IGA) score of clear (0) or almost clear (1) (on a 5-point scale) and a reduction from baseline of >=2 points | At 12 weeks, and 52 weeks after the first treatment
Proportion of Participants Achieving Eczema Area and Severity Index (EASI) Response of >=75 Percent (%) Improvement From Baseline | At week 12 and 52 weeks after the first treatment
Proportion of Participants Achieving >=4 Points improvement in the severity of Pruritus Numerical Rating Scale (NRS) from baseline | At week 12 and 52 weeks after the first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Tower, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451074